CLINICAL TRIAL: NCT02849600
Title: Retrospective Cohort Study of Vital Pulp Therapy in Young Permanent Teeth
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201507090RINC
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Vital Pulp Therapy in Young Permanent Tooth
Keywords: Vital pulp therapy,Young permanent tooth,Treatment outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective cohort study with two specific aims. The first aim focuses on the treatment outcome of different VPT protocols in young permanent tooth. The second aim is to determine if MTA is a suitable material in VPT and related factors potentially influencing prognosis.

DETAILED DESCRIPTION:
Unlike fully developed teeth, the root canal treatment of young permanent teeth is particularly complex and difficult due to its large apical opening, short root length and thin canal wall. In modern endodontics, vital pulp therapy (VPT), a biological based procedures designed to restore functional pulp-dentin complex and promote continued root development, has been considered as an alternative treatment modality. Mineral Trioxide Aggregate (MTA) has been recommended for uses in VPT with preliminary studies, showing promising results. However, lack of high level of evidence trials, inconsistent treatment protocols and follow-up periods, heterogeneous selection criteria, result VPT unreliable and difficult to reach a consensus on the efficacy of MTA. Therefore, we propose this retrospective cohort study with two specific aims. The first aim focuses on the treatment outcome of different VPT protocols in young permanent tooth. The second aim is to determine if MTA is a suitable material in VPT and related factors potentially influencing prognosis. Subjects for the study will be identified from patients who received VPT at the Department of Dentistry in the National Taiwan University Hospital from 1999 to 2014 and have returned for tooth follow up at least one year after treatment. Treatment outcomes will be judged by analyzing clinical and radiographic data, which will be evaluated by 3 independent dentists. The radiographs will be evaluated using a geometrical imaging program-NIH Image J, to calculate the percentage increase in root length and width. Statistical analysis will be applied using the SPSS program to assess the treatment's success rates at the various follow-up periods. The differences will be statistically analyzed performing chi-square test, Fisher exact test, and t-test, using a statistical significance at p<0.05.

ELIGIBILITY:
1. Subjects should be ASA I health person
2. Subject have at least one young permanent tooth received vital pulp therapy, including direct pulp capping, partial pulpotomy, full pulpotomy, partial pulpectomy, apexification and pulp revascularization
3. Subjects have returned for post-treatment clinical and radiographic examination follow up at least one year after treatment

Ages: 7 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The patients who have young permanent tooth and received vital pulp therapy at the Department of Dentistry in the National Taiwan University Hospital from 1999 to 2014 .
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
clinical success | 2 year
  clinical success: no clinical sympton and sign and tooth retained in oral cavity

SECONDARY OUTCOMES:
radiographic success | 2 year
  radiographic success: complete healed of apical lesion, apical foramen closed, root increased in length, root canal wall increased in thickness

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Ling Lee, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No